CLINICAL TRIAL: NCT02486107
Title: Prospective Cohort Study of Outcome After Minimally Invasive Posterior Surgery (Posterior Percutaneous Endoscopic Foraminotomy or Tubular Retractor Assisted Micro-foraminotomy) for Single Level Cervical Foraminal Stenosis
Brief Title: Prospective Cohort Study of Outcome After Minimally Invasive Posterior Cervical Spine Surgery
Acronym: PECD
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Collaborators: Seoul National University Bundang Hospital (Other); Kyungpook National University Hospital (Other)
Responsible Party: Principal Investigator, Chun Kee Chung, professor, Seoul National University Hospital
Other Study IDs: PECD
Record Dates: First submitted 2015-05-20; First posted 2015-07-01 (Estimated); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Spinal Curvature
Keywords: cervical vertebra; surgery; tubular retractor; endoscope
MeSH Terms: conditions — Spinal Curvatures | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- PECD: percutaneous endoscopic cervical foraminotomy
  Interventions: Procedure: surgical procedure
- MTPF: microscopic tubular retractor assisted foraminotomy
  Interventions: Procedure: surgical procedure
- ACDF: anterior cervical discectomy and fusion
  Interventions: Procedure: surgical procedure

INTERVENTIONS:
Procedure: surgical procedure

SUMMARY:
In case of cervical foraminal stenosis without central stenosis, there are several options; anterior discectomy and fusion (ACDF), tubular retractor assisted micro-foraminotomy (MTPF) and posterior percutaneous cervical foraminotomy and discectomy (P-PECD). P-PECD is a modern technique and there was no RCT with MTPF, although P-PECD showed not inferior result to ACDF. Nowadays MTPF and P-PECD are minimally invasive surgical techniques, but there was no comparative study.

The primary object of the study is to compare radiological outcome (segment angle) after MTPF or P-PECD.

DETAILED DESCRIPTION:
P-PECDs are performed in Seoul National University Hospital MTPFs are performed in Kyoung-Pook National University Hospital and ACDF are performed in Seoul National University Bundang Hospital.

ELIGIBILITY:
Inclusion Criteria:

* cervical radicular pain
* no cervical myelopathy

Exclusion Criteria:

* motor weakness less than MMT Gr III
* cervical myelopathy
* OPLL and myelopathy
* previous cervical spine surgery
* combined fracture or spinal tumor

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Alpha = 0.05, Beta = 0.2, q1 = 0.5, effect size = 0.6 drop rate 12% 52 patients in each group
Sampling Method: Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
change of segmental angle | postoperative 1 year

SECONDARY OUTCOMES:
operation time | postoperative 1 year
neck/arm pain | postop 1 year
neck disability, index | postop 1 year
cervical curvature | postop 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Chun Kee Chung, Professor, Principal Investigator — Seoul National University Hospital
Locations (3):
- South Korea (3):
  - Kyoung-Pook National University Hospital, Seoul, Province
  - Seoul National University Bundang Hospital, Seoul
  - Seoul National University Hospital, Seoul